CLINICAL TRIAL: NCT00184600
Title: A 36-month, Multi-centre, Open-label, Randomised, Parallel-group Trial Comparing the Safety, Efficacy and Durability of Adding a Basal Insulin Versus a Twice Daily Insulin Mixture Versus a Meal-time Rapid-Acting Insulin in Subjects With Type 2 Diabetes Inadequately Controlled on Therapy With Oral Agents, and Assessing the Requirement for More Complex Insulin Regimens to Achieve and Maintain Glycaemic Control, Their Efficacy and Durability
Brief Title: Comparison of Insulin Detemir, Insulin Aspart and Biphasic Insulin Aspart 30 With OAD Treatment in Type 2 Diabetes
Acronym: 4T
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1613; 2004-000514-38 (EudraCT Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin detemir (basal insulin) (Experimental): Individually adjusted insulin detemir injected subcutaneously once daily before bed and administered in combination with current OAD treatment. Subjects had the option to add a second pre-breakfast basal insulin analogue injection if pre-breakfast but not pre-dinner meal plasma glucose targets were met. In the second and third years, a second insulin formulation was added if subjects failed to achieve or to maintain good glycaemic control, defined as two consecutive HbA1c measurements exceeding 6.5% or a single measurement exceeding 7.5%. Subjects randomised to insulin detemir once (or twice) daily were asked to add insulin aspart three times daily with meals i.e. a basal-bolus insulin analogue regimen.
  Interventions: Drug: insulin detemir
- Insulin aspart (prandial insulin) (Active Comparator): Individually adjusted insulin aspart injected subcutaneously at meal-times (breakfast, lunch and dinner) and administered in combination with current OAD treatment. In the second and third years, a second insulin formulation was added if subjects failed to achieve or to maintain good glycaemic control, defined as two consecutive HbA1c measurements exceeding 6.5% or a single measurement exceeding 7.5%. Subjects randomised to insulin aspart three times a day with meals were asked to add insulin detemir once or twice daily i.e. a basal-bolus insulin analogue regimen.
  Interventions: Drug: biphasic insulin aspart
- Biphasic insulin aspart 30 (biphasic insulin) (Active Comparator): Individually adjusted biphasic insulin aspart 30 injected subcutaneously twice daily with meals (breakfast and dinner) and administered in combination with current OAD treatment. In the second and third years, a second insulin formulation was added if subjects failed to achieve or to maintain good glycaemic control, defined as two consecutive HbA1c measurements exceeding 6.5% or a single measurement exceeding 7.5%. Subjects randomised to biphasic insulin aspart twice daily were asked to add insulin aspart at lunchtime (midday) i.e. an augmented pre-mixed insulin analogue regimen.
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: biphasic insulin aspart — Treat-to-target (individually adjusted dose), subcutaneously (under the skin) injection, once or twice daily plus option for insulin aspart
  Arms: Insulin aspart (prandial insulin)
Drug: insulin detemir — Treat-to-target (individually adjusted dose), subcutaneously (under the skin) injection, once or twice daily plus option for insulin aspart
  Arms: Insulin detemir (basal insulin)
Drug: insulin aspart — Treat-to-target (individually adjusted dose), subcutaneously (under the skin) injection, twice daily plus option for insulin detemir
  Arms: Biphasic insulin aspart 30 (biphasic insulin)

SUMMARY:
This trial is conducted in Europe.

The aim of this research study is to compare the efficacy (reduction in HbA1c and in blood glucose levels) of insulin detemir, insulin aspart and biphasic insulin aspart 30, when added to current OAD (oral anti-diabetic drug) treatment in subjects with type 2 diabetes and to verify the safety of use (number and severity of episodes of hypoglycaemia, body weight and side effects).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Insulin naive
* On OAD treatment for at least 4 months with metformin, a sulphonylurea or a combination
* Body Mass Index (BMI) below or equal to 40.0 kg/m2
* HbA1c (glycosylated haemoglobin): 7.0%-10% (both inclusive)

Exclusion Criteria:

* Proliferative retinopathy
* Recurrent major hypoglycaemia
* Cardial problems
* Uncontrolled hypertension
* Impaired hepatic or renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2004-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (50):
- Ireland (2):
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Galway
- United Kingdom (48):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Addlestone
  - Novo Nordisk Investigational Site, Airdrie
  - Novo Nordisk Investigational Site, Ashton-under-Lyne
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Berkshire
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Bournemouth
  - Novo Nordisk Investigational Site, Bradford
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Bury St Edmunds
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Colchester
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Crawley
  - Novo Nordisk Investigational Site, Derby
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Gillingham
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Haywards Heath
  - Novo Nordisk Investigational Site, Headington
  - Novo Nordisk Investigational Site, High Wycombe
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Kettering
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, Livingstone
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Middlesbrough
  - Novo Nordisk Investigational Site, Newcastle
  - Novo Nordisk Investigational Site, Norfolk
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Rugby
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Skipton
  - Novo Nordisk Investigational Site, Stevenage
  - Novo Nordisk Investigational Site, Torquay
  - Novo Nordisk Investigational Site, Welwyn Garden City
  - Novo Nordisk Investigational Site, Whiston
  - Novo Nordisk Investigational Site, Wirral, Merseyside

REFERENCES:
- [Result] Holman RR, Farmer AJ, Davies MJ, Levy JC, Darbyshire JL, Keenan JF, Paul SK; 4-T Study Group. Three-year efficacy of complex insulin regimens in type 2 diabetes. N Engl J Med. 2009 Oct 29;361(18):1736-47. doi: 10.1056/NEJMoa0905479. Epub 2009 Oct 22. PMID 19850703
- [Result] Holman RR, Thorne KI, Farmer AJ, Davies MJ, Keenan JF, Paul S, Levy JC; 4-T Study Group. Addition of biphasic, prandial, or basal insulin to oral therapy in type 2 diabetes. N Engl J Med. 2007 Oct 25;357(17):1716-30. doi: 10.1056/NEJMoa075392. Epub 2007 Sep 21. PMID 17890232
- [Result] Jenkins N, Hallowell N, Farmer AJ, Holman RR, Lawton J. Participants' experiences of intensifying insulin therapy during the Treating to Target in Type 2 Diabetes (4-T) trial: qualitative interview study. Diabet Med. 2011 May;28(5):543-8. doi: 10.1111/j.1464-5491.2010.03200.x. PMID 21480965
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 58 sites across the United Kingdom and Ireland. Recruitment period: November 2004-August 2006
Pre-assignment Details: Eligible subjects continued their current oral anti-diabetic drug (OAD) treatment (metformin and/or sulphonylurea) without changing the dose throughout the trial. Subjects were asked not to alter their current diet and activities throughout the trial unless clinically necessary. Subjects fasted from 22:00 the evening prior to randomisation.
Groups:
- Insulin Detemir (Basal Insulin): Individually adjusted insulin detemir injected subcutaneously once daily before bed and administered in combination with current OAD treatment. At week 24 and thereafter, if two consecutive measurements of HbA1c were at least 8%, or one measurement of HbA1c was at least 10% the subject was deemed to have unacceptable hyperglycaemia and a second insulin formulation was added. Subjects had the option to add a second pre-breakfast basal insulin analogue injection if pre-breakfast but not pre-dinner meal plasma glucose targets were met. In the second and third years, a third insulin formulation was added if subjects failed to achieve or to maintain good glycaemic control, defined as two consecutive HbA1c measurements exceeding 6.5% or a single measurement exceeding 7.5%. Subjects randomised to insulin detemir once (or twice) daily were asked to add insulin aspart three times daily with meals i.e. a basal-bolus insulin analogue regimen
- Insulin Aspart (Prandial Insulin): Individually adjusted insulin aspart injected subcutaneously at meal-times (breakfast, lunch and dinner) and administered in combination with current OAD treatment. At week 24 and thereafter, if two consecutive measurements of HbA1c were at least 8%, or one measurement of HbA1c was at least 10% the subject was deemed to have unacceptable hyperglycaemia and a second insulin formulation was added. In the second and third years, a third insulin formulation was added if subjects failed to achieve or to maintain good glycaemic control, defined as two consecutive HbA1c measurements exceeding 6.5% or a single measurement exceeding 7.5%. Subjects randomised to insulin aspart three times a day with meals were asked to add insulin detemir once or twice daily i.e. a basal-bolus insulin analogue regimen
- Biphasic Insulin Aspart 30 (Biphasic Insulin): Individually adjusted biphasic insulin aspart 30 injected subcutaneously twice daily with meals (breakfast and dinner) and administered in combination with current OAD treatment. At week 24 and thereafter, if two consecutive measurements of HbA1c were at least 8%, or one measurement of HbA1c was at least 10% the subject was deemed to have unacceptable hyperglycaemia and a second insulin formulation was added. In the second and third years, a third insulin formulation was added if subjects failed to achieve or to maintain good glycaemic control, defined as two consecutive HbA1c measurements exceeding 6.5% or a single measurement exceeding 7.5%. Subjects randomised to biphasic insulin aspart twice daily were asked to add insulin aspart at lunchtime (midday) i.e. an augmented pre-mixed insulin analogue regimen
Period: Overall Study
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Started | 234 | 239 | 235
Completed | 189 | 188 | 201
Not Completed | 45 | 51 | 34
Not completed — Adverse Event | 9 | 0 | 5
Not completed — Death | 3 | 9 | 7
Not completed — Lack of Efficacy | 3 | 1 | 3
Not completed — Lost to Follow-up | 4 | 6 | 1
Not completed — Protocol Violation | 2 | 2 | 3
Not completed — Withdrawal by Subject | 20 | 28 | 12
Not completed — Unclassified | 4 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin) | Total
Number analyzed (Participants) | 234 | 239 | 235 | 708
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.87 (9.97) | 61.60 (10.54) | 61.67 (8.93) | 61.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 87 | 76 | 254
  Male | 143 | 152 | 159 | 454
Race/Ethnicity, Customized [Number; unit: participants]
  White | 218 | 214 | 221 | 653
  Mixed | 2 | 4 | 1 | 7
  Asian / Asian British | 9 | 15 | 11 | 35
  Black / Black British | 2 | 5 | 2 | 9
  Other | 3 | 1 | 0 | 4
Smoking [Number; unit: participants] — Identifying participants as smokers/non-smokers
  participants
    Non Smoker, Never Smoked | 106 | 88 | 82 | 276
    Ex Smoker | 95 | 108 | 120 | 323
    Current Smoker | 33 | 43 | 33 | 109
Oral Anti-Diabetic Drugs (OADs) [Number; unit: participants] — Identifying which OAD (oral anti-diabetic drug) treatment the participant is on
  participants
    Metformin | 2 | 0 | 4 | 6
    Sulphonylurea | 8 | 12 | 10 | 30
    Metformin + Sulphonylurea | 224 | 227 | 221 | 672
Diabetic complication, Retinopathy [Number; unit: participants] — Diabetic complication at baseline
  participants
    Yes | 43 | 45 | 34 | 122
    No | 191 | 194 | 201 | 586
Diabetic complication, Neuropathy [Number; unit: participants] — Diabetic complication at baseline
  participants
    Yes | 39 | 55 | 41 | 135
    No | 195 | 184 | 194 | 573
Diabetic complication, Nephropathy [Number; unit: participants] — Diabetic complication at baseline
  participants
    Yes | 23 | 24 | 21 | 68
    No | 211 | 215 | 214 | 640
Diabetic complication, Macroaniopathy [Number; unit: participants] — Diabetic complication at baseline
  participants
    Yes | 44 | 42 | 52 | 138
    No | 190 | 197 | 183 | 570
Duration of diabetes [Median (Inter-Quartile Range); unit: years] — Number of years since diagnosis
  years | 9 (5.13) [6 to 12] | 9 (5.54) [6 to 14] | 9 (5.23) [6 to 12] | 9 [6 to 13]
Alcohol [Median (Inter-Quartile Range); unit: units] — Number of units consumed weekly. One unit of alcohol = 10ml pure alcohol by volume or 8g by weight.
  units | 4 (9.16) [2 to 12] | 5 (7.88) [2 to 12] | 6 (9.61) [2 to 12] | 5 [2 to 12]
Weight [Mean (Standard Deviation); unit: kg] — Weight of participants
  kg | 85.52 (16.25) | 84.92 (14.43) | 86.91 (16.82) | 85.8 (15.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI of participants
  kg/m^2 | 29.82 (4.59) | 29.74 (4.51) | 30.34 (4.73) | 29.8 (4.6)
Waist [Mean (Standard Deviation); unit: cm] — Waist circumference of participants
  cm
    Men | 104 (12) | 102 (11) | 104 (12) | 103 (12)
    Women | 97 (12) | 100 (11) | 98 (13) | 98 (12)
Eight-point Capillary Plasma Glucose Profiles [Mean (Standard Deviation); unit: mg/dL]
  All time pointsexcluding 3 am | 196 (43) | 200 (49) | 202 (47) | 200 (47)
  Fasting plasma | 171 (47) | 173 (49) | 175 (50) | 173 (49)
  Postprandial | 223 (50) | 227 (56) | 229 (54) | 227 (54)
  At 3 am | 164 (56) | 164 (59) | 171 (58) | 166 (58)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c (Glycosylated Haemoglobin) at Month 12
Description: HbA1c values offer evidence of the efficacy and durability of the insulin regimens.
Time Frame: Baseline, Month 12
Population: Intention to treat analyses (ITT) included all those randomised. Missing data was imputed by SAS Proc MI (Multiple Imputation), using the non-parametric Propensity Score method for data with monotone missing pattern under the assumption of non-normality and the Bayesian Monte Carlo Markov Chain approach for data with values missing intermittently.
Measure: Mean (Standard Deviation); unit: percentage (%) of total haemoglobin
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
percentage (%) of total haemoglobin
  Baseline | 8.45 (0.80) | 8.55 (0.78) | 8.63 (0.81)
  Month 12 | 7.64 (0.96) | 7.20 (1.06) | 7.33 (0.95)

2. Primary Outcome: HbA1c (Glycosylated Haemoglobin) at Month 36
Description: HbA1c values offer evidence of the efficacy and durability of the insulin regimens.
Time Frame: Baseline, Month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage (%) of total haemoglobin
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
percentage (%) of total haemoglobin
  Baseline | 8.45 (0.80) | 8.55 (0.78) | 8.63 (0.81)
  Month 36 | 7.11 (1.13) | 7.04 (1.17) | 7.22 (1.11)

3. Secondary Outcome: Percentage of Participants (Total Participants and the Subset of Participants Who Did Not Have an Hypoglycaemic Episode) Achieving a Month 12 Value in HbA1c Below or Equal to 6.5%
Description: Two participant counts are listed. The first is the percentage of total participants who achieved the target (HbA1c below or equal to 6.5%) at Month 12. The second is the percentage of subset of participants who achieved the target and did not have either minor or major hypoglycaemic episode within the four weeks prior to the month 12 exam. Minor hypoglycaemic episode is an episode in which the participant was able to treat her/himself and plasma glucose was below 3.1 mmol/L (56 mg/dL). Major hypoglycaemic episode is an episode in which the participant was unable to treat her/himself.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
percentage of participants
  Total participants who achieved target | 8.1 | 23.9 | 17.0
  Subset who achieved target, n=18, 50, 39 | 78.9 | 43.9 | 52.5

4. Secondary Outcome: Percentage of Participants Achieving a Month 36 Value in HbA1c Below or Equal to 6.5%
Description: Percentage of participants who achieved the target (HbA1c below or equal to 6.5%) at Month 36
Time Frame: Month 36
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
percentage of participants | 43.2 | 44.8 | 31.9

5. Secondary Outcome: Number of Hypoglycaemic Events Per Participant Per Year at Month 12 for All Participants and the Subset Who Achieved Target HbA1c Below or Equal to 6.5%
Description: Rate of hypoglycaemic events was calculated as the median number of events per participant per year, defined as grade 1 (symptoms only), 2 (minor) and 3 (major). Symptoms only if self-measured plasma glucose level of 3.1 mmol/L (56 mg/dL) or more. Minor (grade 2) if able to treat her/himself and plasma glucose was below 3.1 mmol/L (56 mg/dL). Major (grade 3) if unable to treat her/himself. Rates are reported for all participants and for the subset of participants who achieved target HbA1c below or equal to 6.5%.
Time Frame: Month 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hypoglycaemic events/participant/year
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
hypoglycaemic events/participant/year
  All participants, Grade 1 | 2.0 [0.0 to 6.0] | 8.0 [3.0 to 19.2] | 5.0 [1.0 to 11.1]
  All participants, Grade 2 | 0 [0 to 2.0] | 8.0 [2.9 to 17.7] | 3.9 [1.0 to 9.0]
  All participants, Grade 3 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  All participants, Grade 2 or 3 | 0 [0 to 2.0] | 8.0 [3.0 to 18.0] | 3.9 [1.0 to 9.0]
  Achieved HbA1c target, Grade 1, n=18, 50, 39 | 3.9 [0 to 5.2] | 7.8 [2.0 to 21.0] | 5.4 [1.5 to 12.8]
  Achieved HbA1c target, Grade 2, n=18, 50, 39 | 3.0 [0 to 4.9] | 8.0 [2.0 to 20.0] | 4.0 [1.5 to 11.4]
  Achieved HbA1c target, Grade 3, n=18, 50, 39 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Achieved HbA1c target, Grade 2 or 3, n=18, 50, 39 | 3.0 [0 to 4.9] | 8.7 [2.9 to 20.0] | 4.0 [1.9 to 11.8]

6. Secondary Outcome: Number of Hypoglycaemic Events Per Participant Per Year at Month 36 for All Participants and the Subset Who Achieved Target HbA1c Below or Equal to 6.5%
Description: as for outcome 5
Time Frame: Month 36
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hypoglycaemic events/participant/year
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
hypoglycaemic events/participant/year
  All participants, Grade 1 | 2.7 [2.3 to 3.0] | 5.7 [4.3 to 7.2] | 3.8 [3.3 to 4.3]
  All participants, Grade 2 | 1.7 [1.3 to 2.0] | 5.5 [4.3 to 6.9] | 3.0 [2.3 to 4.0]
  All participants, Grade 3 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  All participants, Grade 2 or 3 | 1.7 [1.3 to 2.0] | 5.7 [4.3 to 7.0] | 3.0 [2.3 to 4.0]
  Achieved HbA1c target, Grade 1, n=73, 70, 55 | 3.0 [1.7 to 3.7] | 5.7 [3.5 to 7.7] | 3.0 [1.7 to 3.9]
  Achieved HbA1c target, Grade 2, n=73, 70, 55 | 2.0 [1.3 to 2.7] | 5.3 [3.8 to 8.0] | 2.7 [1.7 to 5.2]
  Achieved HbA1c target, Grade 3, n=73, 70, 55 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Achieved HbA1c target, Grade 2 or 3, n=73, 70, 55 | 2.0 [1.3 to 2.7] | 5.5 [4.0 to 8.0] | 3.0 [1.7 to 5.3]

7. Secondary Outcome: Percentage of Participants Who Required A Second Insulin Therapy by Month 12
Description: Percentage of participants who required a second insulin formulation to be added to their treatment. This outcome offers evidence to the efficacy and durability of the insulin regimens.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
percentage of participants | 17.9 | 4.2 | 8.9

8. Secondary Outcome: Percentage of Participants Who Required A Second Insulin Therapy by Month 36
Description: as for outcome 7
Time Frame: Month 36
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
percentage of participants | 89 | 82 | 88

9. Secondary Outcome: Change From Baseline in Body Weight at Month 12
Time Frame: Week 0 (baseline), month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
kilogram | 1.9 (4.2) | 5.7 (4.6) | 4.7 (4.0)

10. Secondary Outcome: Change From Baseline in Body Weight at Month 36
Time Frame: Week 0 (baseline), month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
kilograms | 3.6 (0.5) | 6.4 (0.5) | 5.7 (0.5)

11. Secondary Outcome: Change in Eight-point Capillary Plasma Glucose Profiles (Self-measured) at 12 Months
Description: For each visit and telephone contact, participants were asked to perform in advance three capillary glucose profiles (using blood glucose metre provided for the trial) obtained before breakfast and before the evening meal for participants in the biphasic and basal groups and before meals and two hours after meals and at bedtime in the prandial group.
Time Frame: Baseline, month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
mg/dL
  All timepoints excluding 3am | -43 (43) | -65 (43) | -59 (54)
  Fasting | -59 (52) | -23 (49) | -45 (56)
  Postprandial | -47 (54) | -83 (54) | -68 (63)
  3am | -40 (70) | -34 (59) | -52 (70)

12. Secondary Outcome: Change in Eight-point Capillary Plasma Glucose Profiles (Self-measured) at 36 Months
Description: as for outcome 11
Time Frame: Baseline, month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
mg/dL
  All timepoints excluding 3am | -58 (43) | -67 (47) | -56 (47)
  Fasting | -47 (49) | -49 (45) | -50 (47)
  Postprandial | -67 (50) | -85 (59) | -61 (58)
  3am | -45 (77) | -27 (70) | -38 (77)

13. Secondary Outcome: Quality of Life as Measured by the EuroQol Group 5-Dimension Self-Report Questionnaire Score (EQ5D) at 12 Months
Description: The EuroQol Group 5-Dimension Self-Report Questionnaire score (EQ5D) is a standardised instrument for use as a measure of health outcome in medical research. Responses can be used to generate a single numerical value associated with a given health state. The scale of values is graded from -0.59 to 1.00, with lower scores indicating a poorer health status. A score of 0 represents no quality of life and scores less than 0 represent states perceived by the respondent to be worse than death.
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
units on a scale | 0.78 [0.75 to 0.81] | 0.76 [0.73 to 0.79] | 0.76 [0.73 to 0.80]

14. Secondary Outcome: Quality of Life as Measured by the EuroQol Group 5-Dimension Self-Report Questionnaire Score (EQ5D) at 36 Months
Description: as for outcome 13
Time Frame: Month 36
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
units on a scale | 0.80 [0.77 to 0.83] | 0.77 [0.73 to 0.81] | 0.76 [0.71 to 0.80]

15. Secondary Outcome: Number of Participants Having an 'Other' Adverse Event
Time Frame: Up to month 37 (36 months of treatment plus 1 month follow-up)
Population: Safety population consisting of all randomised participants exposed to at least one dose of trial drug(s).
Measure: Number; unit: participants
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Number analyzed (Participants) | 234 | 239 | 235
participants | 227 | 235 | 228

ADVERSE EVENTS:
Time Frame: The adverse events were collected from the first trial-related activity once the subject had signed the informed consent, up until 28 days after the last clinic visit. Total reporting period for adverse events was 162 weeks.
Description: The safety analysis set contains all randomised subjects exposed to at least one dose of trial drug(s).
Arm/Group | Insulin Detemir (Basal Insulin) | Insulin Aspart (Prandial Insulin) | Biphasic Insulin Aspart 30 (Biphasic Insulin)
Serious Adverse Events (participants affected / at risk) | 78/234 | 79/239 | 105/235
Other Adverse Events (participants affected / at risk) | 227/234 | 235/239 | 228/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (Basal Insulin) (N=234) | Insulin Aspart (Prandial Insulin) (N=239) | Biphasic Insulin Aspart 30 (Biphasic Insulin) (N=235)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 5 (5)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 4 (5) | 2 (4) | 8 (11)
Angina unstable (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial stenosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 1 (1) | 1 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Biopsy liver (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Borderline ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Bronchiectasis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchpulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (5) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 1 (1) | 4 (5)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 6 (6)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3)
Change of bowel habit (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 5 (5) | 1 (6) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 4 (4) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Dislocation of joint prosthesis (General disorders) | 1 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Drug dispensing error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dupuytren's contracture operation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Femoral arterial stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Galbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Graft infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (7) | 13 (13) | 12 (14)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infective exacerbation of chronic obstructive airways (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (4)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Left ventribular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (4)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 6 (6) | 4 (4) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 4 (4) | 2 (2)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 6 (7)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatolithiasis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Penile prosthesis insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (3) | 0 (0)
Pernicious anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Pulse absent (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skull fracture base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Smear cervix abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Stent related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wrong drug administered (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (Basal Insulin) (N=234) | Insulin Aspart (Prandial Insulin) (N=239) | Biphasic Insulin Aspart 30 (Biphasic Insulin) (N=235)
Abdominal discomfort (Gastrointestinal disorders) | 14 (33) | 16 (24) | 27 (40)
Abdominal pain (Gastrointestinal disorders) | 9 (12) | 7 (7) | 14 (20)
Anaemia (Blood and lymphatic system disorders) | 19 (19) | 13 (14) | 14 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (16) | 23 (32) | 25 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (40) | 38 (42) | 28 (35)
Bronchitis (Infections and infestations) | 12 (17) | 10 (13) | 6 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 48 (66) | 51 (63) | 38 (46)
Depression (Psychiatric disorders) | 8 (10) | 12 (12) | 16 (16)
Diabetic retinopathy (Eye disorders) | 19 (20) | 10 (10) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 60 (115) | 53 (75) | 45 (63)
Dizziness (Nervous system disorders) | 20 (28) | 16 (23) | 15 (17)
Dyspepsia (Gastrointestinal disorders) | 21 (38) | 14 (15) | 13 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 20 (24) | 13 (14)
Ear infection (Infections and infestations) | 6 (8) | 11 (15) | 17 (17)
Fall (Injury, poisoning and procedural complications) | 20 (24) | 20 (23) | 16 (20)
Fatigue (General disorders) | 12 (15) | 10 (12) | 4 (7)
Gastroenteritis (Infections and infestations) | 10 (13) | 8 (12) | 14 (15)
Infection (Infections and infestations) | 50 (84) | 55 (88) | 59 (89)
Influenza (Infections and infestations) | 37 (55) | 29 (33) | 33 (43)
Injection site haematoma (General disorders) | 39 (49) | 34 (50) | 34 (46)
Injection site mass (General disorders) | 18 (23) | 7 (7) | 16 (21)
Joint swelling (Musculoskeletal and connective tissue disorders) | 14 (15) | 14 (14) | 8 (8)
Localised infection (Infections and infestations) | 9 (13) | 12 (14) | 16 (20)
Malaise (General disorders) | 15 (38) | 18 (38) | 18 (27)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (14) | 13 (15) | 7 (11)
Nasopharyngitis (Infections and infestations) | 108 (251) | 97 (211) | 99 (208)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 35 (51) | 31 (55) | 27 (37)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 (37) | 31 (35) | 36 (41)
Paraesthesia (Nervous system disorders) | 13 (13) | 11 (16) | 13 (18)
Pharyngitis (Infections and infestations) | 13 (17) | 8 (8) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 11 (14) | 12 (12) | 14 (14)
Upper respiratory tract infection (Infections and infestations) | 33 (51) | 28 (51) | 27 (35)
Urinary tract infection (Infections and infestations) | 32 (67) | 24 (31) | 30 (60)
Viral infection (Infections and infestations) | 12 (12) | 10 (13) | 13 (17)
Vomiting (Gastrointestinal disorders) | 45 (80) | 44 (68) | 43 (71)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones are reached. This includes the right to not release interim results of clinical trials, because that can invalidate results of the entire trial. At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.